CLINICAL TRIAL: NCT05325515
Title: The Effect of Effervescent and Buffered Alendronate on Bone Turnover Compared to Conventional Alendronate: A Randomized Non-inferiority Study
Brief Title: The Effect of Effervescent Alendronate on Bone Turnover
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Torben Harsløf, MD, PhD, consultant in endocrinology, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Binosto_1
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Osteopenia or Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Intervention Model Description: 2 study arms in which participants are allocated by randomization 1:1. Randomixation is performed in 8 blocks of 8.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fosamax (conventional alendronate) (Active Comparator): Conventional alendronate 70mg weekly for 16 weeks
  Interventions: Drug: Conventional alendronate
- Binosto (effervescent and buffered alendronate) (Experimental): Effervescent and buffered alendronate70mg weekly for 16 weeks
  Interventions: Drug: Effervescent and buffered alendronate

INTERVENTIONS:
Drug: Conventional alendronate — Conventional alendronate 70mg weekly
  Arms: Fosamax (conventional alendronate)
Drug: Effervescent and buffered alendronate — Effervescent and buffered alendronate 70mg weekly
  Arms: Binosto (effervescent and buffered alendronate)

SUMMARY:
64 postmenopausal women are randomized to treatment with either effervescent and buffered alendronate or conventional alendronate -both 70mg weekly for 16 weeks to see if bone turnover is suppressed to the same extent as in the conventional formulation with the effervescent form.

DETAILED DESCRIPTION:
Alendronate is mainstay in the treatment of osteoporosis but is often discontinued due to gastro-intestinal side-effects. These side effects are believed to be caused by a low gastric pH induced by the drug. Effervescent and buffered alendronate is a new formulation that increases gastric pH and thereby decreases risk of side effects but the clinical effect of the drug is not fully elucidated. In the present study 64 postmenopausal women with a bone mineral density T-score < -1 are randomized 1:1 to open label treatment with effervescent and buffered alendronate or conventional alendronate 70 mg weekly for 16 weeks. The primary end-point is change in the bone resorption marker "carboxy-terminal collagen crosslinks" from baseline to 16 weeks. The decrease in the two groups is compared using non-inferiority statistics. Secondary end-points include change in the bone formation marker "propeptide of type 1 procollagen", rate of change in the two bone markers and occurence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* 2 years since last menstrual bleeding
* Bone mineral density T-score < -1 at either lumbar spine or hip
* CTx > 0.42 µg/L

Exclusion Criteria:

* Ever treatment for osteoporosis
* Indication for teriparatide treatment
* Treatment with oral systemic glucocorticoids within last 12 months
* Rheumatoid arthritis
* Inflammatory bowel disease
* Untreated thyroid disease
* Primary hyperparathyroidism
* Diabetes mellitus
* eGFR < 60 mL/min
* Cancer within last 2 years except basal cell carcinoma of the skin
* Hormone therapy
* Unstable liver disease
* Contraindications for alendronate
* Major gastrointestinal disease within 12 months (eg. esophagitis, ulcer, major surgery).
* Vitamin D < 50nmol/L

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
CTx | baseline to week 16
  Change in the bone resorption marker CTx

SECONDARY OUTCOMES:
P1NP | baseline to week 16
  Change in the bone resorption marker P1NP

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus C, Central Jutland, Denmark